CLINICAL TRIAL: NCT04774770
Title: HED-Start: A Randomised Controlled Trial to Evaluate a Positive Skills Intervention for Patients New on Haemodialysis
Brief Title: HED-Start: Evaluating a Positive Skills Intervention for Patients New on Haemodialysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Collaborators: National Kidney Foundation, Singapore (Other)
Responsible Party: Principal Investigator, Konstadina Griva, Associate Professor of Health Psychology and Behavioural Medicine, Nanyang Technological University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NKFRC/2018/01/02
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: End Stage Renal Disease on Dialysis; End Stage Renal Failure on Dialysis; End Stage Renal Disease; End Stage Kidney Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Care providers (dialysis nurses) and outcomes assessors (research staff conducting the baseline and follow-up questionnaires) will be blinded to participant allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HED-Start Intervention arm (Experimental): Participants assigned to the intervention arm will undergo 4 sessions of the HED-Start program. Each session is 2 hours long and will be conducted fortnightly.
  Interventions: Behavioral: HED-Start
- Standard care arm (No Intervention): Participants assigned to the standard care arm will proceed with routine standard care.

INTERVENTIONS:
Behavioral: HED-Start — The HED-Start Program is a cognitive-behavioral intervention based on self-management and motivational interviewing principles.
  Arms: HED-Start Intervention arm

SUMMARY:
Hemodialysis patients often experience barriers and misperceptions that hinder adjustment to life on dialysis. This study seeks to explore a group-based intervention (titled HED-Start) developed to improve self-care and emotional wellbeing among incident hemodialysis patients.

DETAILED DESCRIPTION:
There are potentially modifiable psychosocial barriers and misperceptions about life on dialysis that hinder adjustment outcomes. It is hypothesized that these may include: poor understanding on what is needed or 'how to implement treatment principles', misperceptions related to disease and treatment, catastrophizing beliefs about impact of dialysis and low level of confidence on ability to manage treatment regime and renegotiate life roles as a "dialysis patient".

This study seeks to explore the feasibility and acceptability of implementing a two-arm parallel randomized controlled trial of a group-based intervention (titled HED-Start). HED-Start is specifically developed to reduce psychological distress and support self-care and self-management outcomes in incident hemodialysis patients.

Drawing on self-management and motivational interviewing principles paradigm, the HED-Start program aims to facilitate acquisition of skills and knowledge to support and improve self-care and emotional adjustment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with end-stage kidney disease (ESKD) and established on hemodialysis with the National Kidney Foundation Singapore (NKF) for fewer than 90 days
* At least 21 years old
* Proficient in spoken and written English or Mandarin

Exclusion Criteria:

* Unwilling or unable to give informed consent or refuse to be randomized
* Have cognitive impairments or psychiatric conditions that preclude consent
* Are currently involved in other intervention trials
* Are failing on dialysis and approaching end of life (supportive/palliative care pathway)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Anxiety and Depression (HADS) scores from baseline | Participants will be assessed at two time points: [T1] Baseline and [T2] 3 months post-randomization
  Hospital Anxiety and Depression Scale (HADS). The HADS comprises two subscales (anxiety; depression) and can be totaled to produce an overall scale score. Scores range from 0 to 21 for each subscale, and from 0 to 42 for the overall score. Higher scores are indicative of worse anxiety and depression symptoms.

SECONDARY OUTCOMES:
Change in Quality of life (WHOQOL-BREF) scores from baseline | Participants will be assessed at two time points: [T1] Baseline and [T2] 3 months post-randomization
  World Health Organization Quality of Life instrument (WHOQOL-BREF). Two global items (overall quality of life; general health) and two subscales (psychological health; social relationships) from the WHOQOL-BREF are used. Global scores range from 1 to 5, while subscale scores range from 4 to 20. Higher scores indicate better quality of life.
Change in kidney disease-related quality of life (KDQOL-SF) scores from baseline | Participants will be assessed at two time points: [T1] Baseline and [T2] 3 months post-randomization
  Kidney Disease Quality of Life instrument (KDQOL-SF). The Burden of Kidney Disease subscale from the KDQOL-SF will be administered. Scores range from 0 to 100, with a higher score reflecting better quality of life.
Change in Illness Perception scores from baseline | Participants will be assessed at two time points: [T1] Baseline and [T2] 3 months post-randomization
  Brief Illness Perception Questionnaire (BIPQ). The BIPQ consists of 8 subscales (i.e., Consequence, Timeline, Identity, Personal Control, Treatment Control, Concern, Coherence, and Emotional Representation). Subscale scores range from 0 to 10, with higher scores reflective of more negative illness perceptions.
Change in Positive and Negative Affect scores from baseline | Participants will be assessed at two time points: [T1] Baseline and [T2] 3 months post-randomization
  Scale of Positive and Negative Experience (SPANE). The SPANE comprises 6 items assessing positive affect and 6 items assessing negative affect. Subscale scores range from 6 to 30. Higher scores in the Positive and Negative affect subscale indicate greater positive and negative affect respectively.
Change in Self-Efficacy for Managing Chronic Disease 6-item Scale scores from baseline | Participants will be assessed at two time points: [T1] Baseline and [T2] 3 months post-randomization
  Self-Efficacy for Managing Chronic Disease 6-item Scale. The overall scale score ranges from 1 to 10. Higher scores reflect greater self-efficacy.
Change in Benefit finding in hemodialysis (BFS) scores from baseline | Participants will be assessed at two time points: [T1] Baseline and [T2] 3 months post-randomization
  Benefit Finding Scale (BFS). Two subscales (personal growth; acceptance) and an overall score can be computed. All scores range from 1 to 4, with a higher score reflecting a greater extent of benefit finding.
Change in Resilience scores from baseline | Participants will be assessed at two time points: [T1] Baseline and [T2] 3 months post-randomization
  2-item Connor-Davidson Resilience Scale (CD-RISC-2). The CD-RISC-2 score ranges from 0 to 8. Higher scores indicate greater resilience.
Change in Health Education Impact Questionnaire scores from baseline | Participants will be assessed at two time points: [T1] Baseline and [T2] 3 months post-randomization
  Health Education Impact Questionnaire (heiQ). Six subscales from the heiQ (Positive and Active Engagement in Life, Skill and Technique Acquisition, Constructive Attitudes and Approaches, Self-Monitoring and Insight, Health Services Navigation, and Social Integration and Support) will be used to assess other self-management skills. Scores range from 1 to 4. Higher scores indicate greater proficiency with the relevant skill domain.

CONTACTS AND LOCATIONS:
Overall Officials: Konstadina Griva, PhD, Principal Investigator — Nanyang Technological University
Locations (1):
- National Kidney Foundation Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes
All deidentified IPD that underlie results in a publication will be available upon reasonable request.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Griva K, Chia JMX, Goh ZZS, Wong YP, Loei J, Thach TQ, Chua WB, Khan BA. Effectiveness of a brief positive skills intervention to improve psychological adjustment in patients with end-stage kidney disease newly initiated on haemodialysis: protocol for a randomised controlled trial (HED-Start). BMJ Open. 2021 Sep 21;11(9):e053588. doi: 10.1136/bmjopen-2021-053588. PMID 34548369